CLINICAL TRIAL: NCT00831246
Title: Prevention of Post-Op Ileus After Gynecologic Surgery Using Chewing Gum
Brief Title: Prevention of Ileus After Gynecologic Surgery Using Chewing Gum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aultman Health Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2008.03.27.E2; 2008 JMC
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Ileus
Keywords: Ileus,; Gynecologic surgery,; Post-operative,; Flatus
MeSH Terms: conditions — Ileus; Flatulence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients are given standard post-op care with clear liquid diet as tolerated plus chewing gum q8 for 30minute chewing intervals.
  Interventions: Other: chewing gum - Extra Winterfresh
- 2 (Sham Comparator): Patients are given standard post-op care with clear liquid diet as tolerated .
  Interventions: Other: Standard Post-Op Care

INTERVENTIONS:
Other: chewing gum - Extra Winterfresh — Patients are given standard post-op care with clear liquid diet as tolerated plus chewing gum q8 for 30minute chewing intervals.
  Arms: 1
Other: Standard Post-Op Care — Patients are given standard post-op care with clear liquid diet as tolerated.
  Arms: 2

SUMMARY:
This study will attempt to determine if the use of chewing gum can cause the early return of bowel function after gynecologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* All female patients 18 years of age or older undergoing surgery for any gynecologic procedure which the peritoneum is entered and general anesthesia is administered.
* Disease State will not affect inclusion in the study. Women with previous surgeries or other medical conditions will be included as will those undergoing an initial operation.

Exclusion Criteria:

* Patient deemed legally incompetent to sign their own consent
* Women under the age of 18
* Patients lacking their own or a false set of teeth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Incidence of ileus | Until ileus formation or first flatus post-op

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hopkins, MD, Study Chair — Aultman Health Foundation; James M Clark, MD, Principal Investigator — Aultman Health Foundation
Locations (1):
- Aultman Health Foundation, Canton, Ohio, United States